CLINICAL TRIAL: NCT01098877
Title: A Double Blind, Randomized, Placebo Controlled, Dose Escalation Study To Investigate The Pharmacokinetics (In The Fed And Fasted State), Safety And Toleration Of Single Oral Doses Of PF-04634817 In Healthy Volunteers
Brief Title: First In Human Study Of Increasing Oral Doses Of PF-04634817
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B1261002
Record Dates: First submitted 2010-03-26; First posted 2010-04-05 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: Phase1; pharmacokinetics; safety; toleration; pharmacodynamics
MeSH Terms: interventions — PF-04634817

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (11):
- Placebo (Placebo Comparator)
  Interventions: Drug: PF-04634817 Placebo
- Cohort 1, 1mg (Experimental)
  Interventions: Drug: PF-04634817
- Cohort 1, 3mg (Experimental)
  Interventions: Drug: PF-04634817
- Cohort 1, 10mg (Experimental)
  Interventions: Drug: PF-04634817
- Cohort 2, 30mg (Experimental)
  Interventions: Drug: PF-04634817
- Cohort 2, 100mg (Experimental)
  Interventions: Drug: PF-04634817
- Cohort 2, 300mg (Experimental)
  Interventions: Drug: PF-04634817
- Cohort 3, 600mg (Experimental)
  Interventions: Drug: PF-04634817
- Cohort 3, 900mg (Experimental)
  Interventions: Drug: PF-04634817
- Cohort 3, up to 900mg (fed) (Experimental)
  Interventions: Drug: PF-04634817
- Cohort 3, placebo (fed) (Placebo Comparator)
  Interventions: Drug: PF-04634817 Placebo

INTERVENTIONS:
Drug: PF-04634817 Placebo — Oral solution, placebo, single dose
  Arms: Placebo
Drug: PF-04634817 — Oral solution, 1mg, single dose
  Arms: Cohort 1, 1mg
Drug: PF-04634817 — Oral solution, 3mg, single dose
  Arms: Cohort 1, 3mg
Drug: PF-04634817 — Oral solution, 10mg, single dose
  Arms: Cohort 1, 10mg
Drug: PF-04634817 — Oral solution, 30mg, single dose
  Arms: Cohort 2, 30mg
Drug: PF-04634817 — Oral solution, 100mg, single dose
  Arms: Cohort 2, 100mg
Drug: PF-04634817 — Oral solution, 300mg, single dose
  Arms: Cohort 2, 300mg
Drug: PF-04634817 — Oral solution, 600mg, single dose
  Arms: Cohort 3, 600mg
Drug: PF-04634817 — Oral solution, 900mg, single dose
  Arms: Cohort 3, 900mg
Drug: PF-04634817 — Oral solution, up to 900mg, single dose after food
  Arms: Cohort 3, up to 900mg (fed)
Drug: PF-04634817 Placebo — Oral solution, placebo, single dose after food
  Arms: Cohort 3, placebo (fed)

SUMMARY:
The study will evaluate the hypothesis that at doses and plasma concentrations which affect pharmacodynamic markers of activity at the chemokine receptors, CCR2 and CCR5, the compound is safe and well tolerated. It will also evaluate the hypothesis that the pharmacokinetic profile is robust and consistent with a once or twice a day therapeutic administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female (of non-child bearing potential) subjects between 18 and 55 years of age.
* Body mass index of 17.5 to 30.5 kg/m2 and total body weight > 50kg.

Exclusion Criteria:

* Evidence or history of any clinically significant disease.
* Treatment with an investigational drug within 30 days of study start
* Use of prescription and non-prescription medicines within 7 days of study start

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety and toleration: adverse events, supine and standing vital sign measurements, telemetry, 12-lead ECGs, blood and urine tests | 0-3 days
Plasma pharmacokinetics: Cmax, Tmax, AUClast, AUCinf, AUC0-24, CL/F, Vz/F and T1/2 | 0-4 days
Urinary pharmacokinetics: Aet (mount excreted in urine), Aet% and CLr | 0-2 days
p-ERK inhibition in human monocytes | 0-3 days
Change in circulating monocytes | 0-3 days

SECONDARY OUTCOMES:
Change from baseline in plasma MCP-1 | 0-3 days
MIP 1B stimulated CCR5 receptor internalization | 0-3 days
MCP-1 stimulated CCR5 receptor internalization | 0-3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1261002&StudyName=First%20In%20Human%20Study%20Of%20Increasing%20Oral%20Doses%20Of%20PF-04634817